CLINICAL TRIAL: NCT02816866
Title: Comparing Two Modes of Survivorship Care: A Randomized Trial
Brief Title: Comparing Two Modes of Survivorship Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 1007007080; 119700-RSGHP-10-107-01-CPHPS (Other Grant/Funding Number: American Cancer Society)
Record Dates: First submitted 2016-06-17; First posted 2016-06-29 (Estimated); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Childhood Cancer
Keywords: survivorship care; health services; barriers
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- empowered primary care model (Experimental): patients receive an individualized "prescription" for survivorship care prepared by a cancer survivor specialist to be implemented by the primary care doctor
  Interventions: Other: empowered primary care model
- specialty survivor clinic (Experimental): patient attends a specialty survivor clinic at Yale for survivorship care
  Interventions: Other: specialty survivor clinic

INTERVENTIONS:
Other: empowered primary care model — mode of survivorship care
  Arms: empowered primary care model
Other: specialty survivor clinic — mode of survivorship care
  Arms: specialty survivor clinic

SUMMARY:
The main purpose of this study is to research the comparative effectiveness of two potential models of health care to deliver preventive services and chronic care management to the growing population of adult and pediatric survivors of childhood cancer. The central hypothesis is that survivorship care delivered by a subject's primary care doctor after the subject is empowered with individualized follow-up recommendations prepared by a cancer survivor specialist is similar to care provided in a specialty survival clinic.

DETAILED DESCRIPTION:
Although 80% of children with cancer will be cured of their primary disease, at least 70% of survivors will develop chronic medical, neurocognitive, and/or emotional conditions as a complication of their therapy. Most of these conditions are amenable to prevention and early intervention. In response, the Institute of Medicine strongly advised that all cancer patients should receive survivorship care with the following key elements: 1) a summary of previous cancer therapy, 2) individualized life-long screening for potential adverse therapy-related effects, and 3) education regarding desirable health behaviors. However, less than 30% of survivors receive recommended care. There is a tremendous need for research that addresses how to best implement evidence-based recommendations for this population.

Two main health care delivery models have been advocated for survivorship care, but no comparison studies exist. The first model is a specialty survivor clinic, usually at a cancer treatment center. The second model, termed the empowered primary care model, involves patients receiving an individualized "prescription" for follow-up care prepared by a cancer survivor specialist to be implemented by the primary care doctor. Each model poses unique strengths and weaknesses. Specialty survivor clinics can be expensive and geographically inaccessible, can cause anxiety and stress to patients, and can accommodate limited numbers of patients. Primary care doctors may lack adequate expertise and time for these complex patients. Unless we know how these approaches compare with regard to quality of care and risks, advocates and policy makers will be stymied in their efforts to support the health needs of cancer survivors. This study seeks to compare subjects randomized to the empowered primary care model vs. a specialty survivor clinic.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of any malignancy at age <18 years and reported to Yale-New Haven Hospital or Connecticut Children's Medical Center (CCMC) tumor registry
* Currently alive and cancer-free
* Primary residence within approximately 100 miles of Yale-New Haven Hospital or CCMC
* ≥ 1 year status post completion of all cancer-related therapy
* Elapsed time of less than 12.0 years since diagnosis of malignancy
* Speaking and writing knowledge of English. For subjects <18 years, at least one parent must satisfy this requirement.
* No previous attendance at the Yale HEROS or CCMC Reach for the STARS survivorship clinics, or other specialty survivorship clinic

Exclusion Criteria:

* n/a

Ages: 1 Year to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 106 (Actual)
Dates: Start 2010-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
adherence to guideline-recommended surveillance (medical record abstraction) | 12 months post-intervention
  quality of survivorship care
number of newly-identified late effects of therapy (medical record abstraction) | 12 months post-intervention
  quality of survivorship care

SECONDARY OUTCOMES:
anxiety (Brief Symptom Inventory (BSI)) | 12 months post-intervention
  adverse effects of receiving survivorship care
depression (Behavior Assessment System for Children, 2nd Edition (BASC-2)) | 12 months post-intervention
  adverse effects of receiving survivorship care
post-traumatic stress symptoms (Post-Traumatic Stress Disorder Reaction Index (PTSD-RI)) | 12 months post-intervention
  adverse effects of receiving survivorship care
level of physical activity (2008 questionnaires of the Behavioral Risk Factor Surveillance System (BRFSS)) | 12 months post-intervention
  adherence to desirable health behaviors
avoidance of tobacco (2008 questionnaires of the Behavioral Risk Factor Surveillance System (BRFSS)) | 12 months post-intervention
  adherence to desirable health behaviors
intake of at least five servings per day of fruits and vegetables (2008 questionnaires of the Behavioral Risk Factor Surveillance System (BRFSS)) | 12 months post-intervention
  adherence to desirable health behaviors

CONTACTS AND LOCATIONS:
Overall Officials: Nina S Kadan-Lottick, MD, MSPH, Principal Investigator — Yale University

IPD SHARING:
Plan to Share IPD: No